CLINICAL TRIAL: NCT00004448
Title: Alternate Day Prednisone or Daily Fish Oil Supplements in Patients With Immunoglobulin A Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Southwest Pediatric Nephrology Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/13463; R01DK049368 (NIH); SPNSG-94.052 (Other: Southwest Pediatric Nephrology Study Group)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2008-09

CONDITIONS: IgA Glomerulonephritis
Keywords: IgA glomerulonephritis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Glomerulonephritis, IGA; Rare Diseases; Urogenital Diseases | interventions — Fatty Acids, Omega-3; Omacor; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prednisone (Experimental): Tapering regimen of alternate-day prednisone tablets (Deltasone)
  Interventions: Drug: prednisone
- omega-3 fatty acids (Experimental): Omega 3 fatty acid Omacor
  Interventions: Drug: omega-3 fatty acids
- Placebo (Placebo Comparator): Placebo for prednisone or fatty acid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: omega-3 fatty acids
  Other Names: Omacor
  Arms: omega-3 fatty acids
Drug: prednisone
  Other Names: Deltasone
  Arms: Prednisone
Drug: Placebo
  Arms: Placebo

SUMMARY:
OBJECTIVES:

Evaluate the efficacy of alternate day prednisone versus daily fish oil supplements in slowing or preventing the decline in renal function in children, adolescents, and young adults with moderate to severe immunoglobulin A nephropathy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is randomized, double blind, placebo controlled, multicenter study.

Patients are randomized into one of three treatment arms: placebo, prednisone, or fish oil. The placebo arm is further randomized to receive either fish oil placebo capsules or prednisone placebo tablets.

Arm I: Patients receive placebo tablets or capsules for 2 years. Arm II: Patients receive a tapering regimen of prednisone tablets administered every other day for 2 years in the absence of unacceptable toxicity.

Arm III: Patients receive fish oil capsules daily for 2 years. Patients may also receive enalapril for hypertension. Patients are followed every 3 months for 3 years after treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically confirmed immunoglobulin A nephropathy (IgAN) Patients must have either: - Persistent severe proteinuria alone (urine Pr/Cr ratio at least 1.0) OR - Moderate proteinuria plus renal biopsy changes indicating risk of progression (glomerulosclerosis or proliferation) --Prior/Concurrent Therapy-- Endocrine therapy: At least 1 month since any prior prednisone No more than 3 months of prior prednisone therapy since renal biopsy Other: At least 1 month since any prior immunosuppressive therapy or fish oils No more than 3 months of prior immunosuppressive therapy or fish oil administration since renal biopsy --Patient Characteristics-- Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) AST less than 2 times ULN No known chronic liver disease Renal: Protein excretion greater than 0.5 g/1.73 m2/24 hours OR Urine protein/creatinine ratio greater than 0.5 on 2 occasions at least 4 weeks apart in the 6 months prior to study Creatinine clearance at least 50 mL/min Other: No systemic lupus erythematosus No Henoch-Schonlein purpura No diabetes mellitus, cataracts, aseptic necrosis of any bone, or other conditions potentially exacerbated by prednisone therapy Not pregnant Adequate contraception required of all fertile patients

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 1997-11 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to failure | Up to 5 years after randomization
  Time to failure was defined as the interval until the eGFR fell to <60% of baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hogg, Study Chair — Southwest Pediatric Nephrology Study Group
Locations (1):
- Medical City Dallas Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Hogg RJ. A randomized, placebo-controlled, multicenter trial evaluating alternate-day prednisone and fish oil supplements in young patients with immunoglobulin A nephropathy. Scientific Planning Committee of the IgA Nephropathy Study. Am J Kidney Dis. 1995 Nov;26(5):792-6. doi: 10.1016/0272-6386(95)90445-x. No abstract available. PMID 7485134
- [Result] Hogg RJ, Lee J, Nardelli N, Julian BA, Cattran D, Waldo B, Wyatt R, Jennette JC, Sibley R, Hyland K, Fitzgibbons L, Hirschman G, Donadio JV Jr, Holub BJ; Southwest Pediatric Nephrology Study Group. Clinical trial to evaluate omega-3 fatty acids and alternate day prednisone in patients with IgA nephropathy: report from the Southwest Pediatric Nephrology Study Group. Clin J Am Soc Nephrol. 2006 May;1(3):467-74. doi: 10.2215/CJN.01020905. Epub 2006 Apr 12. PMID 17699247
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639